CLINICAL TRIAL: NCT04544501
Title: A Randomized Controlled Trial to Enhance the Use of Genetic Counseling and Testing in Latinas
Brief Title: Enhance the Use of Genetic Counseling and Testing in Latinas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: Basser Center for BRCA (Unknown); Nueva Vida, Inc. (Industry); Capital Breast Care Center (Unknown); Virginia Commonwealth University (Other); Arlington Free Clinic (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00001436
Record Dates: First submitted 2020-06-18; First posted 2020-09-10 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2021-12

CONDITIONS: Hereditary Breast and Ovarian Cancer Syndrome
Keywords: Latinas; Intervention
MeSH Terms: conditions — Hereditary Breast and Ovarian Cancer Syndrome

STUDY DESIGN:
Intervention Model Description: 28 Latina women at risk for HBOC will be randomly assigned to one arm after completing the baseline assessment.
  We will conduct a Hybrid Type 1 design to (1) test the effectiveness of two intervention approaches (video vs. FORCE fact sheet) in enhancing GCRA uptake and psychosocial outcomes and to (2) collect data on implementation outcomes regarding the interventions (video vs. FORCE fact sheet) and the implementation of a short screening survey to identify at-risk women.
  Given the hybrid design, we will also conduct focus groups with clinic staff, in which we estimate 32 staff to participate. Given their participation in the focus groups, clinic staff are also considered participants, but they are not part of the randomized trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culturally-Targeted Video (Experimental)
  Interventions: Behavioral: Culturally-Targeted Video
- FORCE Fact Sheet (Active Comparator)
  Interventions: Other: FORCE Fact Sheet

INTERVENTIONS:
Behavioral: Culturally-Targeted Video — Culturally targeted narrative video: "Is My Cancer Hereditary? Rosa Visits a Genetic Counselor." With R03 funding (R03CA191543) we developed a culturally targeted narrative video for at-risk Latinas. A multidisciplinary team of researchers collaborated with filmmakers to develop the script and video. The script was informed by health behavior conceptual models, evidence-based risk communication strategies, and formative research (40 interviews with providers and at-risk Latinas). The script addressed identified knowledge gaps (e.g., incorrect belief that pap smears screen for ovarian cancer), facilitators (e.g., inform family cancer risk), barriers (e.g., emotional concerns), and cultural factors (e.g., respect). The 18-minute video illustrates the GCRA process with the story of Rosa, a Latina cancer survivor at increased risk of HBOC. Rosa learns about HBOC risk factors, overcomes barriers, and attends genetic counseling.
  Arms: Culturally-Targeted Video
Other: FORCE Fact Sheet — A publically available Spanish-language fact sheet about HBOC and GCRA developed by FORCE.
  Arms: FORCE Fact Sheet

SUMMARY:
The investigators will conduct a two-arm RCT to evaluate the preliminary effectiveness of a culturally-adapted video developed by the team vs. a FORCE fact sheet on enhancing genetic cancer risk assessment (GCRA; including genetic counseling and option for genetic testing) uptake and psychosocial outcomes among Latinas at increased risk for hereditary breast and ovarian cancer (HBOC).

DETAILED DESCRIPTION:
The investigators will conduct a two-arm RCT to evaluate the preliminary effectiveness of a culturally-adapted video developed by the team vs. FORCE fact sheet on enhancing genetic cancer risk assessment (GCRA; including genetic counseling and option for genetic testing) uptake and psychosocial outcomes among Latinas at increased risk for hereditary breast and ovarian cancer (HBOC).

All participants will receive referrals to free telephone genetic counseling in Spanish to address cost, pragmatic, and language barriers. The investigators will recruit 28 Latina women at-risk of HBOC (14 randomized at each arm) at three sites with sizable Latinx populations. The sites include community clinics/health organizations and hospitals with whom we have established collaborations [Georgetown University (DC); Virginia Commonwealth University (VA)].

Results will improve efforts to translate genomic guidelines into practice and will reduce disparities by evaluating a low cost highly disseminable culturally-targeted video while gathering data on effectiveness and implementation.

Aim 1. Evaluate the impact of video vs. FORCE fact sheet on GCRA and testing uptake and psychosocial outcomes.

Aim 2. Assess implementation potential and needs by evaluating feasibility, acceptability, reach, and adoption of the intervention arms (video and FORCE fact sheet) and of the HBOC screening process at the community clinics.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years-old
* Self-identify as Latina
* Fluent in Spanish
* Meet NCCN criteria for breast and/or ovarian genetic cancer risk assessment based on -personal or family history of cancer
* Have not received genetic counseling or genetic testing
* Able to provide informed consent
* No other members of the same family have participated
* Must have access to the internet via smartphone, computer, or another device.

Exclusion Criteria:

* Not fluent in Spanish
* Previously received genetic counseling or genetic testing for HBOC
* Previously participated in another interventional study about HBOC and GCRA

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Genetic counseling uptake | Baseline survey to three months after baseline
  Proportion of participants that receive genetic counseling. The outcome will be assessed by self-report (e.g., Have you received genetic counseling in the past three months?) and confirmed with the genetic counseling company records.

SECONDARY OUTCOMES:
Genetic testing uptake | Baseline survey to three months after baseline
  Proportion of participants that receive genetic testing. The outcome will be assessed by self-report (e.g., Have you received genetic testing in the past three months?) and confirmed with the genetic counseling company records.

OTHER OUTCOMES:
Breast cancer genetics knowledge | Change from baseline to two weeks after baseline and change from baseline to three months after baseline
  Change in knowledge about HBOC and GCRA. Knowledge will be measured using a 13-item Erblich et al., 2005 scale about genetic knowledge about breast cancer. The scale has statements to which participants respond True, False, or I don't Know. The scale is scored based on the accuracy of responses. A higher score indicates higher knowledge. Scores range from 0-13.
Intentions to participate in genetic counseling and genetic testing | Baseline to two weeks after baseline
  Change in intentions to participate in genetic counseling and genetic testing. A 2-item scale developed by Sussner, Jandorf, Thompson, and Valdimarsdottir, 2010 will be used to assess intentions to participate in genetic counseling and testing. Participants respond to a Likert-trype scale from 1 (Not at all) to 5 (Very) how likely it is that they will participate in genetic counseling and testing in the next three months.
Beliefs and attitudes about genetic counseling and genetic testing | Baseline to two weeks after baseline
  Changes in beliefs and attitudes about genetic counseling and genetic testing. The outcome will be assessed by a 30-item scale developed by Sussner, Jandorf, Thompson et al., 2012 in which participants respond to a Likert-type scale from 1 (completely disagree) to 7 (complete agree).
Anticipatory Emotions | Baseline to two weeks after baseline
  Changes in anticipatory emotions about receive genetic counseling. Assessed by participants' responses to how they feel 'right now' about the specific behavior of receiving genetic counseling and testing in the next three months. Responses are in a 7-point Likert-type form (from 1-strongly disagree to 7-strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Alejandra Hurtado de Mendoza, Ph.D, Principal Investigator — Georgetown University
Locations (4):
- United States (4):
  - Capital Breast Care Center, Washington D.C., District of Columbia
  - Nueva Vida, Alexandria, Virginia
  - Arlington Free Clinic, Arlington, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No